CLINICAL TRIAL: NCT00941525
Title: Central Corneal Thickness and 24-hour Fluctuation of Intraocular Pressure
Acronym: CCT-IOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Fotis Topouzis, Professior, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 83155; EudraCT: 2008-004629-41
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
Keywords: Central corneal thickness; 24hour fluctuation of intraocular pressure; Open angle glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ocular hypertensives (Other): This study includes two groups.
  1. Subjects with ocular hypertension and
  2. Controls. Group 2 undergoes only 1 visit (visit 1) without any intervention. Group 1 undergoes visit 1 without intervention. Then they receive treatment (1 eyedrop of latanoprost (0.005%) dosed once a day in both eyes at 8:00pm for a 4-weeks period for 1 month) and undergo the visit 2 under the effect of treatment.
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost — 1 eyedrop of latanoprost (0.005%) dosed once a day at 8:00pm for a 4-weeks period
  Other Names: 0.005% Xalatan

SUMMARY:
The purpose of this study is to determine whether 24-hour fluctuation of intraocular pressure (IOP) is associated with central corneal thickness (CCT) in subjects with ocular hypertension or open angle glaucoma and in age-matched controls. Also to evaluate whether mean IOP reduction as a response to latanoprost (0.005% Xalatan) is associated with CCT, after a 4-weeks period of treatment.

Also, to evaluate whether 24-hour fluctuation of IOP is associated with corneal hysteresis (CH) measured by Ocular Response Analyzer (ORA).

ELIGIBILITY:
Inclusion Criteria:

Males and females >50 years old with:

* Primary Open-Angle Glaucoma newly diagnosed or with anti-glaucoma medical treatment < =12 weeks
* Pseudoexfoliative Glaucoma newly diagnosed or with anti-glaucoma medical treatment <= 12 weeks
* Ocular Hypertensives newly diagnosed or with anti-glaucoma medical treatment <= 12 weeks
* Age-matched controls
* IOP>=22mmHg at the eligibility visit for glaucoma patients and ocular hypertensives

Exclusion Criteria:

For Eye

* Use of any ophthalmic medication (drops) during the study (except for natural tears)
* Inflammation of any aetiology
* Previous eye surgery or laser
* Corneal abnormalities (oedema, dystrophies etc) For Subjects
* Systemic diseases which affect the cornea (such as autoimmune diseases)
* Inability to participate due to advanced age or serious illness
* Mean IOP>36mmHg in either eye at the eligibility visit.
* Subjects who cannot safety discontinue use of all IOP-lowering medication(s) for washout
* Subjects with severe central visual field loss in either eye. Severe central visual field loss is defined as sensitivity <=10dB in at least 2 of the 4 visual field test points closest to the point of fixation
* Other types of glaucoma (such as angle-closure glaucoma and secondary glaucomas)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Correlation analyses between mean central corneal thickness (CCT) and 24-hour intraocular pressure (IOP) fluctuation and between mean CCT and mean IOP reduction from baseline after a 4-weeks period of treatment with latanoprost. | Before and after a 4-weeks period of treatment with latanoprost.

SECONDARY OUTCOMES:
Correlation analyses between corneal hysteresis (CH) and 24-hour intraocular pressure (IOP) fluctuation and between CH and mean IOP reduction from baseline after a 4-weeks period of treatment with latanoprost. | Before and after a 4-weeks period of treatment with latanoprost.

CONTACTS AND LOCATIONS:
Overall Officials: Fotis Topouzis, MD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- A' Department of Ophthalmology, Aristotle University of Thessaloniki, AHEPA Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Nouri-Mahdavi K, Hoffman D, Coleman AL, Liu G, Li G, Gaasterland D, Caprioli J; Advanced Glaucoma Intervention Study. Predictive factors for glaucomatous visual field progression in the Advanced Glaucoma Intervention Study. Ophthalmology. 2004 Sep;111(9):1627-35. doi: 10.1016/j.ophtha.2004.02.017. PMID 15350314
- [Background] Asrani S, Zeimer R, Wilensky J, Gieser D, Vitale S, Lindenmuth K. Large diurnal fluctuations in intraocular pressure are an independent risk factor in patients with glaucoma. J Glaucoma. 2000 Apr;9(2):134-42. doi: 10.1097/00061198-200004000-00002. PMID 10782622
- [Background] European Glaucoma Prevention Study (EGPS) Group; Miglior S, Pfeiffer N, Torri V, Zeyen T, Cunha-Vaz J, Adamsons I. Predictive factors for open-angle glaucoma among patients with ocular hypertension in the European Glaucoma Prevention Study. Ophthalmology. 2007 Jan;114(1):3-9. doi: 10.1016/j.ophtha.2006.05.075. Epub 2006 Oct 27. PMID 17070596
- [Background] Gordon MO, Beiser JA, Brandt JD, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Kass MA. The Ocular Hypertension Treatment Study: baseline factors that predict the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):714-20; discussion 829-30. doi: 10.1001/archopht.120.6.714. PMID 12049575
- [Background] Orzalesi N, Rossetti L, Invernizzi T, Bottoli A, Autelitano A. Effect of timolol, latanoprost, and dorzolamide on circadian IOP in glaucoma or ocular hypertension. Invest Ophthalmol Vis Sci. 2000 Aug;41(9):2566-73. PMID 10937568
- [Background] Larsson LI, Mishima HK, Takamatsu M, Orzalesi N, Rossetti L. The effect of latanoprost on circadian intraocular pressure. Surv Ophthalmol. 2002 Aug;47 Suppl 1:S90-6. doi: 10.1016/s0039-6257(02)00296-5. PMID 12204704
- [Background] Orzalesi N, Rossetti L, Bottoli A, Fumagalli E, Fogagnolo P. The effect of latanoprost, brimonidine, and a fixed combination of timolol and dorzolamide on circadian intraocular pressure in patients with glaucoma or ocular hypertension. Arch Ophthalmol. 2003 Apr;121(4):453-7. doi: 10.1001/archopht.121.4.453. PMID 12695241
- [Background] Liu JH, Kripke DF, Weinreb RN. Comparison of the nocturnal effects of once-daily timolol and latanoprost on intraocular pressure. Am J Ophthalmol. 2004 Sep;138(3):389-95. doi: 10.1016/j.ajo.2004.04.022. PMID 15364220
- [Background] Orzalesi N, Rossetti L, Bottoli A, Fogagnolo P. Comparison of the effects of latanoprost, travoprost, and bimatoprost on circadian intraocular pressure in patients with glaucoma or ocular hypertension. Ophthalmology. 2006 Feb;113(2):239-46. doi: 10.1016/j.ophtha.2005.10.045. PMID 16458092
- [Background] Luce DA. Determining in vivo biomechanical properties of the cornea with an ocular response analyzer. J Cataract Refract Surg. 2005 Jan;31(1):156-62. doi: 10.1016/j.jcrs.2004.10.044. PMID 15721708
- [Background] Congdon NG, Broman AT, Bandeen-Roche K, Grover D, Quigley HA. Central corneal thickness and corneal hysteresis associated with glaucoma damage. Am J Ophthalmol. 2006 May;141(5):868-75. doi: 10.1016/j.ajo.2005.12.007. Epub 2006 Mar 9. PMID 16527231
- [Background] Kotecha A, Elsheikh A, Roberts CR, Zhu H, Garway-Heath DF. Corneal thickness- and age-related biomechanical properties of the cornea measured with the ocular response analyzer. Invest Ophthalmol Vis Sci. 2006 Dec;47(12):5337-47. doi: 10.1167/iovs.06-0557. PMID 17122122
- [Background] Larsson LI. Intraocular pressure over 24 hours after repeated administration of latanoprost 0.005% or timolol gel-forming solution 0.5% in patients with ocular hypertension. Ophthalmology. 2001 Aug;108(8):1439-44. doi: 10.1016/s0161-6420(01)00605-4. PMID 11470697
- [Background] Kida T, Liu JH, Weinreb RN. Effect of 24-hour corneal biomechanical changes on intraocular pressure measurement. Invest Ophthalmol Vis Sci. 2006 Oct;47(10):4422-6. doi: 10.1167/iovs.06-0507. PMID 17003435